CLINICAL TRIAL: NCT02888353
Title: An Expanded Evaluation of the Safety of Clinically Indicated Magnetic Resonance Imaging (MRI) in Patients With Pacemakers and Implanted Cardioverter Defibrillators
Brief Title: Magnetic Resonance Imaging (MRI) in Patients With Pacemakers and Implanted Cardioverter Defibrillators
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00068447
Record Dates: First submitted 2015-12-28; First posted 2016-09-05 (Estimated); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Device:MRI
Keywords: Magnetic Resonance Imaging and Pacemakers ICD

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Device: MRI no pre-screen (Experimental): Clinically Indicated MRI will be done in patients with cardiac devices (pacemakers and defibrillators).
  Patients will not be pre-screened prior to hospital visit.
  Interventions: Device: Device: MRI

INTERVENTIONS:
Device: Device: MRI — Perform MRI in patients with cardiac devices

SUMMARY:
Ferromagnetic Implants such as permanent pacemakers (PPM's) and Implantable Cardioverter Defibrillators (ICD's) have traditionally been accepted as contraindications to Magnetic Resonance Imaging (MRI) due to safety concerns. Over the past several years, MRI safety has been established in patients with pacemakers or ICD's but only in patients in whom strict vetting procedures were implemented. These vetting procedures were initially developed to eliminate devices, leads and device/lead circumstances thought to carry increased risk. Over recent years however, objective scientific evidence has failed to support this concern raising the question as to whether or not these vetting procedures are necessary.

Investigators hypothesize that in view of the existing objective scientific data, evolution of device technology and the fact that the investigators have scanned more than 2,000 devices safely (RPN03-08-11-12 and 00051707) ICD's and pacemakers and device circumstances previously excluded from MRI protocols can be safely scanned without prior vetting.

This is a prospective, non randomized, cohort study. Seventeen Hundred participants with an implanted ICD or pacemaker and a clinical need for MRI will be included in the study. Unlike previous studies where strict vetting procedures were implemented pre-procedure, All patients with a pacemaker or ICD and clinical need for an MRI will be eligible for inclusion in the study provided participants meet standard MRI inclusion/exclusion safety criteria.

DETAILED DESCRIPTION:
Pilot studies of approximately 1500 patients, RPN #03-08-12-11 and 00051707 (manuscript submitted) demonstrated the safety of most contemporary implanted rhythm management devices in the MRI environment given appropriate precautions.

When pilot studies were developed, there was a theoretical concern that there may be an increased risk associated with some device and device circumstances including: 1) PPM's or leads implanted prior to 1996; 2) ICD's implanted prior to 2000; 3) abandoned or endocardial leads; 4) leads implanted <6 weeks; 5) ICD's where patient is pacemaker dependent.

While it was reasonable to be hyper vigilant when initiating pilot studies by including restrictive inclusion criteria, the natural evolution of the devices and device related technologies coupled with a lack of objective scientific data to support investigator's early safety concerns has caused investigators to reevaluate their necessity. For example, older pacemakers and ICD's that previously excluded potential participants are now obsolete; all have expired batteries and have been explanted. Similarly, the technological evolution of ICD's includes ICD's that are now capable of providing ongoing asynchronous pacing including in the MRI environment. Despite some concern that abandoned, epicardial and newly implanted leads may be at increased risk of heating or subject to torque, when investigators evaluated 15 participants with these lead issues and exposed them to MRI (off protocol in life threatening situations) there were no adverse problems seen.

The vetting procedures investigators implemented in pilot studies required that a registered nurse obtain all patient device information and chest xrays (when indicated) from referring physicians, review them in advance of allowing participants to schedule an MRI, and exclude any patient who did not meet inclusion criteria. Investigators found that these procedures were time consuming and expensive (as they required a part time Registered Nurse (RN) salary). In addition, in some cases, patients who might have derived considerable benefit from an MRI were excluded from obtaining one and the time it took to adhere to the vetting procedures needlessly delayed the MRI in some participants, causing them unnecessary stress and frustration and even adversely affecting their clinical care.

MRI's will be done in participants who require a clinically indicated MRI without implementing the vetting procedures investigators included in pilot studies. Participants with implanted pacemakers and ICD's will only be eligible for MRI at Johns Hopkins Hospital (JHH) if they agree to participate in this study. All studies will be done in the 1.5 Tesla MRI unit. Since the first 100 participants were scanned in investigator's initial protocol 03-08-11-12, MRI scan sequences, field intensity and fields of exposure have been given no special consideration given the presence of the pacemaker or ICD and there have been no adverse or unanticipated problems. For this reason, investigators do not feel it is necessary to impose any special restrictions (related to field intensity or scan sequences/exposure) in this protocol. In the event that any device manufacturer indicates the need for including additional safety precautions investigators will amend the protocol immediately to include them.

Electrocardiogram (ECG) monitoring pads will be placed on the patient for the duration of the study. Heart rate, blood pressure, O2 saturation will be monitored non-invasively throughout the study by a registered electrophysiology nurse who is Advanced Cardiac Life Support (ACLS )certified, fully trained in cardiac device management and familiar with the research protocol as well as the implications of scanning patients with cardiac devices. In addition to the electrophysiology nurse, two fully certified MRI technologists familiar with scanning participants with implanted devices will be present in the control room the entire time the participant is scanned. The scanner is located in close proximity to the electrophysiology laboratory where Electrophysiology physicians perform procedures, hence at all times at least one, but typically more than one Electrophysiology physician who knows both the participant and the MRI device procedure will be available. A Zoll external defibrillator with transthoracic pacing capabilities, ACLS drugs and a fully equipped crash cart will be readily available at all times in an area that is adjacent to the MRI control room.

Prior to the MRI, participants will be handed an alarm button and instructed to notify the MRI technologist if for any reason he/she feels it is necessary and particularly in the event that any unusual pains or sensations are experienced. Participants can be seen by the technologist and the nurse who is monitoring the scan through a large window that separates the scanner from the control room. In addition, the MRI technologist frequently initiates conversation between sequences by asking the patient; "how are you".

All devices will undergo a complete interrogation and testing prior to imaging and following imaging. PPMs will be programmed to an asynchronous mode if dependent and to an inhibited mode in patients without pacemaker dependence.

The pacemaker function of ICD's in pacemaker independent patients will be programmed to ventricular inhibited (VVI) mode at 50 bpm. Pacemaker dependent participants with ICD's who were previously excluded from prior studies will no longer be excluded as ICD's are now reliably capable of maintaining adequate pacing when programmed to an asynchronous pacing mode..

After the appropriate MRI protocol for each MRI patient is completed, the device will be re-programmed to its original settings and completely interrogated and retested to detect any changes in device performance.

All MRI's are clinically indicated and therefore standard of care. The participants participation in the study will terminate when they complete a 1-6 week follow-up device evaluation that will also be done as standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Patients implanted an ICD or pacemaker who have a clinical need for MR imaging

Exclusion Criteria:

* Patients who complete the MRI standard screening form and are deemed inappropriate for MRI for any reason

Ages: 9 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4500 (Estimated)
Dates: Start 2015-12 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
acute patient safety and device malfunction | 1 hour
  Number of participants with >30% change pre vs. post MRI in each of the following (pacing volts, sensing amplitude, battery life, and impedance (ohms), as a measure of safety

SECONDARY OUTCOMES:
chronic patient safety and device malfunction | 1 to 6 weeks
  Number of participants with >30% change in each of the following (pacing volts, sensing amplitude, battery life, and impedance (ohms) 1 to 6 weeks post MRI as a measure of safety

CONTACTS AND LOCATIONS:
Overall Officials: Henry R Halperin, MD/MA, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Zayed 5 MRI, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Nazarian S, Hansford R, Rahsepar AA, Weltin V, McVeigh D, Gucuk Ipek E, Kwan A, Berger RD, Calkins H, Lardo AC, Kraut MA, Kamel IR, Zimmerman SL, Halperin HR. Safety of Magnetic Resonance Imaging in Patients with Cardiac Devices. N Engl J Med. 2017 Dec 28;377(26):2555-2564. doi: 10.1056/NEJMoa1604267. PMID 29281579
- [Result] Ra J, Oberdier MT, Suzuki M, Vaidya D, Liu Y, Hansford R, McVeigh D, Weltin V, Tao S, Thiemann DR, Nazarian S, Halperin HR. Implantable Defibrillator System Shock Function, Mortality, and Cause of Death After Magnetic Resonance Imaging. Ann Intern Med. 2023 Mar;176(3):289-297. doi: 10.7326/M22-2653. Epub 2023 Jan 31. PMID 36716451
- See also: PubMed Citation #1 — https://pubmed.ncbi.nlm.nih.gov/29281579/
- See also: PubMed Citation #2 — https://pubmed.ncbi.nlm.nih.gov/36716451/